CLINICAL TRIAL: NCT04293185
Title: A Phase 3 Study Evaluating Gene Therapy by Transplantation of Autologous CD34+ Stem Cells Transduced Ex Vivo With the BB305 Lentiviral Vector in Subjects With Sickle Cell Disease
Brief Title: A Study Evaluating Gene Therapy With BB305 Lentiviral Vector in Sickle Cell Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGB-210
Record Dates: First submitted 2020-02-12; First posted 2020-03-03 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — lyfgenia; Excipients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- bb1111 (Experimental): Subjects will receive treatment with a single dose of Drug Product manufactured with autologous CD34+ hematopoietic stem cells collected by plerixafor mobilization and apheresis, transduced with BB305 lentiviral vector (LVV) encoding the human beta-A-T87Q globin gene.
  Plerixafor mobilization and apheresis will also be used for collection of rescue cells.
  Interventions: Genetic: bb1111

INTERVENTIONS:
Genetic: bb1111 — Drug Product is administered by IV infusion following myeloablative conditioning with busulfan.
  Other Names: lovotibeglogene autotemcel; lovo-cel; LentiGlobin BB305 Drug Product for SCD; autologous CD34+ cell-enriched population from patients with SCD that contains HSCs transduced with BB305 LVV encoding the βA-T87Q-globin gene, suspended in cryopreservation solution

SUMMARY:
This is a non-randomized, open-label, multi-site, single-dose, Phase 3 study in approximately 35 adults and pediatric subjects ≥2 and ≤50 years of age with sickle cell disease (SCD). The study will evaluate hematopoietic stem cell (HSC) transplantation (HSCT) using bb1111 (also known as LentiGlobin BB305 Drug Product for SCD).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of SCD, with either βS/βS, βS/β0, or βS/β+ genotype.
* Be ≥2 and ≤50 years of age at time of consent.
* Weigh a minimum of 6 kg.
* Have a Karnofsky performance status of ≥60 (≥16 years of age) or a Lansky performance status of ≥60 (<16 years of age).
* Be treated and followed for at least the past 24 months prior to Informed Consent in medical center(s) that maintained detailed records on sickle cell disease history.
* In the setting of appropriate supportive care measures (e.g., pain management plan), have experienced at least 4 protocol-defined VOEs in the 24 months prior to informed consent.
* Have either experienced HU failure at any point in the past or must have intolerance to HU (intolerance is defined as the patient being unable to continue to take HU per PI judgment).
* Female and male subjects of childbearing potential agree to use 1 method of highly effective contraception from Screening to at least 6 months after drug product infusion.
* Provision of written informed consent for this study by subject, or as applicable, subject's parent(s)/legal guardian(s).

Exclusion Criteria:

* Subjects for whom allogeneic hematopoietic stem cell transplantation (allo-HSCT) is medically appropriate per PI judgment and a willing, human leukocyte antigen (HLA)-matched related hematopoietic stem cell donor is available.
* Severe cerebral vasculopathy, defined by any history of overt ischemic or hemorrhagic stroke, a history of abnormal transcranial Doppler (TCD) or TCD imaging (TCDI) for subjects ≤ 16 years of age (e.g. TCD velocity >200 cm/sec) requiring ongoing chronic transfusions, a Screening TCD or TCDI velocity > 200 cm/sec (central read), a Screening MRA showing > 50% stenosis or occlusion in the circle of Willis (central read), or a Screening MRA showing the presence of Moyamoya (central read).
* Positive for presence of human immunodeficiency virus type 1 or 2 (HIV-1 or HIV-2), hepatitis B, hepatitis C, human T-lymphotropic virus-1 (HTLV-1), active syphilis.
* Clinically significant, active bacterial, viral, fungal, or parasitic infection
* Advanced liver disease, such as

  1. clear evidence of liver cirrhosis, active hepatitis or significant fibrosis (based on MRI or liver biopsy)
  2. liver iron concentration ≥15 mg/g unless liver biopsy shows no evidence of cirrhosis, active hepatitis or significant fibrosis
* Inadequate bone marrow function, as defined by an absolute neutrophil count of <1×10^9/L (<0.5×10^9/L for subjects on hydroxyurea treatment) or a platelet count <100×10^9/L.
* Any contraindications to the use of plerixafor during the mobilization of hematopoietic stem cells and any contraindications to the use of busulfan and any other medicinal products required during the myeloablative conditioning, including hypersensitivity to the active substances or to any of the excipients.
* Patients needing therapeutic anticoagulation treatment during the period of conditioning through platelet engraftment
* Unable to receive pRBC transfusion.
* Prior receipt of an allogeneic transplant.
* Prior receipt of gene therapy.
* Any prior or current malignancy or immunodeficiency disorder, except previously treated, non-life threatening, cured tumors such as squamous cell carcinoma of the skin.
* Immediate family member with a known or suspected Familial Cancer Syndrome.
* Female subject is breastfeeding, pregnant or will attempt to become pregnant from Screening to at least 6 months after drug product infusion.
* Any other condition that would render the subject ineligible for HSCT.
* Participation in another clinical study with an investigational drug within 30 days of screening.
* Presence of a chromosomal abnormality or genetic mutation that may put the subject at an increased risk of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) per Investigator's judgment.
* Presence of genetic mutations that result in the inactivation of 2 or more α-globin genes

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
VOE-CR | 6-18 months post-transplant
  Proportion of subjects achieving complete resolution of VOEs between 6 months and 18 months after drug product infusion

SECONDARY OUTCOMES:
sVOE-CR | 6-18 months post-transplant
  Proportion of subjects achieving complete resolution of severe vaso-occlusive events, between 6 months and 18 months after drug product infusion
Proportion of subjects achieving Globin Response | 6-24 months post-transplant
  Globin Response, defined as meeting the following criteria for a continuous period of at least 6 months after drug product infusion:
  1. Weighted average HbAT87Q percentage of non-transfused total Hb* ≥30% AND
  2. Weighted average non-transfused total Hb* increase of ≥3 g/dL compared to baseline total Hb* OR weighted average non-transfused total Hb* ≥10 g/dL
     * non-transfused total Hb is the total g/dL of HbS + HbF + HbA2 + HbAT87Q
Change in the annualized number of VOEs in the 24 months after drug product infusion compared to the 24 months prior to Informed Consent | 1-24 months post-transplant
Change in the annualized number of severe VOEs in the 24 months after drug product infusion compared to the 24 months prior to Informed Consent. | 1-24 months post-transplant
VOE-CR24 | 6-24 months post-transplant
  Proportion of subjects achieving complete resolution of VOEs between 6 months and 24 months after drug product infusion
sVOE-CR24 | 6-24 months post-transplant
  Proportion of subjects achieving complete resolution of severe VOEs between 6 months and 24 months after drug product infusion
sVOE-75 | 1-24 months post-transplant
  Proportion of subjects achieving at least a 75% reduction in annualized severe VOEs in the 24 months after drug product administration compared to the 24 months prior to Informed Consent.
Weighted average non-transfused total Hb | Month 6, 12, 18 and 24 post-transplant
Weighted average HbS percentage of non-transfused total Hb | Month 6, 12, 18 and 24 post-transplant
Weighted average HbS percentage of non-transfused total Hb ≤70%, ≤60%, ≤50% | Month 6, 12, 18 and 24 post-transplant
Weighted average HbAT87Q percentage of non-transfused total Hb | Month 6, 12, 18 and 24 post-transplant
Weighted average non-HbS percentage of non-transfused total Hb | Month 6, 12, 18 and 24 post-transplant
Average and median of non-transfused total Hb | 1-24 months post-transplant
Average and median of HbS percentage of non-transfused total Hb | 1-24 months post-transplant
Average and median of HbAT87Q percentage of non-transfused total Hb | 1-24 months post-transplant
Average and median of non-HbS percentage of non-transfused total Hb | 1-24 months post-transplant
Change from baseline in absolute reticulocyte count | 1-24 months post-transplant
Change from baseline in percent reticulocytes | 1-24 months post-transplant
Change from baseline in percent erythrocytes | 1-24 months post-transplant
Change from baseline in total bilirubin | 1-24 months post-transplant
Change from baseline in haptoglobin | 1-24 months post-transplant
Change from baseline in lactate dehydrogenase | 1-24 months post-transplant
Change from baseline in ferritin | 1-24 months post-transplant
Change from baseline in liver iron content | 1-24 months post-transplant
Change from baseline in cardiac iron content (if assessed at baseline) | 1-24 months post-transplant
Change from baseline in erythropoietin | 1-24 months post-transplant
Change from baseline in serum transferrin receptor | 1 - 24 months post-transplant
Change from baseline in annualized frequency of packed red blood cell (pRBC) transfusions | 6-24 months post-transplant
Change from baseline in annualized volume of pRBC transfusions | 6-24 months post-transplant
Change from baseline in TCD velocity at Month 12 and Month 24 (for subjects ≤ 16 years old at Informed Consent) | Month 12 and Month 24 post-transplant
Change from baseline in meters walked during the 6-minute walk test | 1 - 24 months post-transplant
Change from baseline in annualized number of SCD-related hospital admissions | 1 - 24 months post-transplant
Change from baseline in annualized number of total days hospitalized | 1 - 24 months post-transplant
Change from baseline in patient-reported quality of life, as measured by PROMIS-57 Version 2.1 for subjects ≥ 18 years of age and PROMIS Pediatric Profile/Parent Proxy Profile 49 Version 2.0 for subjects < 18 years of age | 1 - 24 months post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Anjulika Chawla, MD, FAAP, Study Director — bluebird bio, Inc.
Locations (9):
- United States (9):
  - University of Alabama, Birmingham, Alabama
  - Children's National Hospital, Washington D.C., District of Columbia
  - Tufts Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - Virginia Commonwealth University (VCU), Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Bluebird bio is committed to transparency and appropriately de-identified patient-level datasets and supporting documents may be shared upon completion of study participation and following attainment of applicable marketing approvals associated with this study and consistent with criteria established by bluebird bio and/or industry best practices to maintain the privacy of study participants. For enquiries, please contact us at datasharing@bluebirdbio.com.